CLINICAL TRIAL: NCT05610267
Title: A Retrospective Analysis of the Use of Gentrix® Surgical Matrix for Soft Tissue Reinforcement in Ventral Hernia Repair
Brief Title: Gentrix® Surgical Matrix for Soft Tissue Reinforcement in Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: T-GENVIH-002
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Retrospective chart review — The retrospective chart review will include the full consecutive series of patients between 22 years and 80 years old who underwent abdominal wall reconstruction for achart hernia with Integra Gentrix® Surgical Matrix during the time period between November 1, 2017, and present (90 days prior to the start of data collection).

SUMMARY:
The purpose of this study is to collect additional safety data and demonstrate the performance of Integra Gentrix® Surgical Matrix for reinforcement of ventral hernia repairs.

DETAILED DESCRIPTION:
Retrospective data will be collected and assessed for early post-operative surgical site events and complications in the immediate post-operative period of 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 22 years and 80 years old (inclusive) at time they underwent abdominal wall reconstruction utilizing Gentrix® Surgical Matrix as a reinforcement graft during the time period between November 1, 2017, and present (90 days prior to the start of the data collection)..
2. Subject underwent abdominal wall reconstruction for a hernia(s) using Integra® Gentrix® Surgical Matrix.

Exclusion Criteria:

1. Subject has known allergy to porcine-derived products.
2. Subject required use of Gentrix® device and a second non-Gentrix surgical mesh in the same plane or in different planes for single hernia e.g., Gentrix sublay and a synthetic device in the onlay position.
3. Subject had active necrotizing fasciitis or any current known uncontrolled systemic infection.
4. Subject had uncontrolled diabetes, defined as Hb1AC value >7% within 12 weeks prior to index procedure.
5. Subject has been diagnosed with cirrhosis and/or ascites.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 22 years and 80 years old (inclusive) at time they underwent abdominal wall reconstruction utilizing Gentrix® Surgical Matrix as a reinforcement graft during the time period between November 1, 2017, and present (90 days prior to the start of the data collection).
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Young, MD, Study Director — Integra LifeSciences Corporation
Locations (1):
- Surgical Healing Arts Center, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The retrospective chart review including the full consecutive series of patients between 22 years and 80 years old who underwent abdominal wall reconstruction for a chart hernia with Integra Gentrix® Surgical Matrix during the time period between November 1, 2017, and September 1, 2022 (90 days prior to the start of data collection) started in November 2022 and ended in december 2022. The enrollment occured at a single Surgical center.
Pre-assignment Details: 29 subjects screened, 1 subject, screened failure. 28 subjects, male and female were enrolled and completed the study.
Groups:
- Device: Retrospective Chart Review: Subject has undergone abdominal wall reconstruction for a chart hernia with Integra Gentrix® Surgical Matrix.
Period: Overall Study
Arm/Group | Device: Retrospective Chart Review
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subject has undergone abdominal wall reconstruction for a hernia with Integra Gentrix® Surgical Matrix.
Groups:
- Device: Retrospective Chart Review: Subject has undergone abdominal wall reconstruction for a hernia with Integra Gentrix® Surgical Matrix.
Arm/Group | Device: Retrospective Chart Review
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 21
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post-operative Complications Requiring Procedural Intervention Within 90 Days Post Index Procedure
Description: Percentage of subjects with a post-operative complications requiring procedural intervention within 90 days post index procedure
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Retrospective Chart Review
Number analyzed (Participants) | 28
Participants | 2

2. Secondary Outcome: Incidence of Early Post-operative Complications (Surgical Site Occurrences (SSOs)) Within 90 Days Post Index Procedure
Description: Percentage of subjects with an early post-operative complications (Surgical Site Occurrences (SSOs)) within 90 days post index procedure
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Retrospective Chart Review
Number analyzed (Participants) | 28
Participants | 8

3. Secondary Outcome: Incidence of Surgical Site Infections (SSIs) Post Index Procedure
Description: Percentage of subjects with Surgical Site Infections (SSIs) Post index procedure
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Retrospective Chart Review
Number analyzed (Participants) | 28
Participants | 4

4. Secondary Outcome: Incidence of Later Post-operative Complications After 90 Days Post Index Procedure
Description: Percentage of subjects with a later post-operative complications after 90 days post index procedure
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Retrospective Chart Review
Number analyzed (Participants) | 28
Participants | 4

5. Secondary Outcome: Incidence of Hernia Recurrence Confirmed by Clinical Assessment
Description: Percentage of subjects with a hernia recurrence confirmed by clinical assessment
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Retrospective Chart Review
Number analyzed (Participants) | 28
Participants | 1

6. Secondary Outcome: Incidence of Reoperation Requirement Due to Index Repair
Description: Percentage of subjects with a reoperation requirement due to index repair
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Retrospective Chart Review
Number analyzed (Participants) | 28
Participants | 4

7. Other Pre Specified Outcome: Average Length of Hospital Stay (LOS) Post Index Procedure (Measured in Days)
Description: Number of days between the date of the index procedure and the date of the hospital discharge
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Device: Retrospective Chart Review
Number analyzed (Participants) | 28
Days | 2.8 (2.55)

8. Other Pre Specified Outcome: Rate of Opioid Usage Following Procedure Determined by % of Prescriptions Filled and Refilled
Description: Number of subjects who used opioids following the procedure based on the concomitants medication
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Retrospective Chart Review
Number analyzed (Participants) | 28
Participants | 24

ADVERSE EVENTS:
Time Frame: Retrospective chart review of AEs that occurred between Index Surgery and last follow-up visit up to 14 months
Description: Adverse Event information were collected on any adverse event that the subject experienced between Index Surgery and last follow-up visit up to 14 months.
Arm/Group | Device: Retrospective Chart Review
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 3/28
Other Adverse Events (participants affected / at risk) | 13/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: Retrospective Chart Review (N=28)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1) — Eroded abdominal wall mesh and volvulus of small intestine adhered to the eroded mesh, surgically treatedEroded abdominal wall mesh and volvulus of small intestine adhered to the eroded mesh, surgically treated
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) — Fall originated a different hernia incarcerated abdominal preperitoneal fat pad
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 (1) — Admitted in hospital, adhesions released, obstruction resolved.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: Retrospective Chart Review (N=28)
Intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Application site haematoma (General disorders) | 2 (2)
Instillation site haematoma (General disorders) | 1 (1)
Abdominal wall abscess (Injury, poisoning and procedural complications) | 1 (1)
Abdominal wall infection (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 5 (5)
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 4 (4)
Abscess drainage (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT05610267/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT05610267/SAP_001.pdf